CLINICAL TRIAL: NCT00474903
Title: Randomized, Double-Blinded Phase II Trial of Esomeprazole Versus Esomeprazole + Two Doses of Aspirin in Barrett's Esophagus Patients
Brief Title: Esomeprazole Magnesium With or Without Aspirin in Preventing Esophageal Cancer in Patients With Barrett Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCI-2009-00838; NCI-2009-00838 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAY04-4-01; CDR0000544180; MAYO-MAY04-4-01 (Other: Mayo Clinic); MAY04-4-01 (Other: DCP); N01CN35000 (NIH)
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-01

CONDITIONS: Barrett Esophagus; Esophageal Cancer
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Aspirin; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Arm I (placebo, esomeprazole magnesium) (Active Comparator): Patients receive two oral placebos once daily and oral esomeprazole magnesium (40 mg, twice daily).
  Interventions: Drug: esomeprazole magnesium; Other: placebo
- Arm II (low-dose aspirin, esomeprazole magnesium) (Experimental): Patients receive both an oral placebo and acetylsalicylic acid (81 mg dose), once daily and oral esomeprazole magnesium (40 mg, twice daily).
  Interventions: Drug: acetylsalicylic acid; Drug: esomeprazole magnesium; Other: placebo
- Arm III (higher-dose aspirin, esomeprazole magnesium) (Experimental): Patients receive both an oral placebo and acetylsalicylic acid (325 mg dose), once daily and oral esomeprazole magnesium (40 mg, twice daily).
  Interventions: Drug: acetylsalicylic acid; Drug: esomeprazole magnesium; Other: placebo

INTERVENTIONS:
Drug: acetylsalicylic acid — Given orally
  Arms: Arm II (low-dose aspirin, esomeprazole magnesium); Arm III (higher-dose aspirin, esomeprazole magnesium)
Drug: esomeprazole magnesium — Given orally
Other: placebo — Given orally

SUMMARY:
This randomized phase II trial is studying the effect of esomeprazole magnesium and aspirin on tissue PGE2 levels compared with esomeprazole and placebo. This type of chemoprevention treatment investigates the use of certain drugs to assess whether they assist in the prevention of cancer. The use of esomeprazole magnesium with or without aspirin may help prevent esophageal cancer in patients with Barrett esophagus.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the effects of a 28 day intervention with aspirin 81 mg placebo orally (PO) once daily (QD) + aspirin 325 mg placebo PO QD + esomeprazole 40 mg PO BID versus aspirin 81 mg PO QD + aspirin 325 mg placebo PO QD + esomeprazole 40 mg PO BID versus aspirin 325 mg PO QD + aspirin 81 mg placebo PO QD + esomeprazole 40 mg PO BID on the absolute change in tissue prostaglandin E2 (PGE2) concentration, as determined from Barrett's esophagus mucosal biopsy samples obtained pre- and post-intervention (i.e. two pair-wise comparisons of two different doses of active aspirin regimens versus aspirin placebo group), Specifically, the two active aspirin + esomeprazole arms will be independently analyzed to see if they significantly reduce the mean tissue PGE2 concentration from Pre- to Post-intervention as compared to the aspirin placebo + esomeprazole arm.

SECONDARY OBJECTIVES:

I. To determine if the change in the tissue PGE2 concentration decreases significantly in the aspirin placebo + esomeprazole arm.

II. To compare the change in mean tissue PGE2 concentration between the two active intervention arms to determine which one appears the most promising for further testing.

III. To assess the effects of the three agents (arms) with respect to proliferation (Ki-67), apoptosis (caspase-3 expression), COX-2 expression, and p16 methylation using Pre- and Post-Intervention biopsy samples obtained from Barrett's mucosal tissue.

IV. To evaluate all adverse events associated with each of the three intervention arms.

V. To provide exploratory summaries of PGE2 concentration values by patient subgroups of interest.

VI. To provide descriptive summaries of the esophagogastroduodenoscopy (EGD) results, the rate of dysplasia, adverse events, and the Run-In Agent compliance on all participants that signed a consent form and started the Run-In phase of the trial.

VII. To establish a biospecimen repository archive for future correlative studies.

OUTLINE: This is a multicenter, randomized, double-blind, placebo-controlled study. Patients are stratified according to dysplasia status, gender, and length of Barrett segment of circumferential involvement (5 cm vs = 5 cm). Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive two oral placebos once daily and oral esomeprazole magnesium twice daily.

ARM II: Patients receive oral acetylsalicylic acid (aspirin) and oral placebo once daily and oral esomeprazole magnesium twice daily.

ARM III: Patients receive a higher-dose of oral aspirin (higher than in arm II) and a lower-dose of oral placebo (lower than in arm II) once daily and oral esomeprazole magnesium twice daily.

In all arms, treatment continues for 28 days in the absence of unacceptable toxicity. Tissue samples are collected before and after treatment and examined for tissue-based biomarkers (i.e., PGE_2, Ki-67, caspase-3 apoptosis, and cyclooxygenase-2) by immunohistochemistry, enzyme immunoassay, Western blot, and polymerase chain reaction.

After completion of study therapy, patients are followed 7 - 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Barrett esophagus, meeting all of the following criteria:

  * Presence of specialized columnar epithelium anywhere in the tubular esophagus with ≥ 2 cm of circumferential involvement
  * No evidence of high-grade dysplasia or cancer by esophagogastroduodenoscopy (EGD)
  * No prior histologically confirmed esophageal dysplasia, including cancer
* Adequate Barrett mucosa, defined as ≥ 4 of 8 research samples with≥ 50% intestinal metaplasia in research biopsies
* No ulcer, erosion, plaque, nodule, stricture, or other luminal irregularity within the Barrett's segment or erosive esophagitis (Los Angeles classification > grade A) detected at pre-intervention EGD exam
* Eastern Cooperative Group (ECOG) performance status 0-2
* Hemoglobin normal
* Platelet count ≥ 100,000/mm³
* Aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 2.5 times ULN
* Creatinine ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No nasal polyps associated with asthma or induced or exacerbated by aspirin
* No malignancy within the past 5 years except for nonmelanoma skin cancer
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to the study agents or rescue medication
* No history of endoscopically or radiographically diagnosed peptic ulcer disease (bleeding or nonbleeding)
* No other uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Bleeding disorder
  * Vitamin K deficiency
  * Alcohol abuse (defined as ingestion of ≥ 3 drinks per day)
  * Psychiatric illness or social situations that would limit study compliance
* At least 3 months since prior chronic use (defined as ≥ 7 days during the 3 months preceding the beginning of the Run-in phase) of acetylsalicylic acid (aspirin), nonsteroidal antiinflammatory drug (NSAIDs), or selective cyclooxygenase (COX-2) inhibitors
* At least 3 months since prior investigational agents except innocuous agents with no known interaction with the study agents (e.g., standard dose multivitamins or topical agents for limited skin conditions)
* No prior fundoplication, bariatric surgery, or any other major upper gastrointestinal surgery

  * Prior cholecystectomy allowed
* No other concurrent NSAIDs (including aspirin) or selective COX-2 inhibitor therapy
* No concurrent anticoagulant drugs including, but not limited to, any of the following:

  * Warfarin
  * Heparin
  * Low-molecular weight heparin
  * Clopidogrel bisulfate
  * Extended-release dipyridamole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-04; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Limburg, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Falk GW, Buttar NS, Foster NR, Ziegler KL, Demars CJ, Romero Y, Marcon NE, Schnell T, Corley DA, Sharma P, Cruz-Correa MR, Hur C, Fleischer DE, Chak A, Devault KR, Weinberg DS, Della'Zanna G, Richmond E, Smyrk TC, Mandrekar SJ, Limburg PJ; Cancer Prevention Network. A combination of esomeprazole and aspirin reduces tissue concentrations of prostaglandin E(2) in patients with Barrett's esophagus. Gastroenterology. 2012 Oct;143(4):917-26.e1. doi: 10.1053/j.gastro.2012.06.044. Epub 2012 Jul 11. PMID 22796132

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 122 patients were randomized. Two patients withdrew due to an inadequate number of biopsies and a finding of high-grade dysplasia. Six participants were not evaluable for the primary endpoint due to sample-related issues (e.g., improper temperature, lost or delayed samples), leaving 114 evaluable participants for the primary endpoint.
Pre-assignment Details: Of the 120 participants in the intervention cohort, 114 were evaluable for the primary endpoint (n = 29, 42, and 43 in Arm I, Arm II, and Arm III, respectively).
Groups:
- Arm I (Placebo, Esomeprazole Magnesium): Patients receive two oral placebos once daily and oral esomeprazole magnesium (40 mg, twice daily).
  esomeprazole magnesium: Given orally placebo: Given orally
- Arm II (Low-dose Aspirin, Placebo, Esomeprazole Magnesium): Patients receive both an oral placebo and acetylsalicylic acid (81 mg dose), once daily and oral esomeprazole magnesium (40 mg, twice daily).
  acetylsalicylic acid: Given orally esomeprazole magnesium: Given orally placebo: Given orally
- Arm III (Higher-dose Aspirin, Palcebo, Esomeprazole Magnesium): Patients receive both an oral placebo and acetylsalicylic acid (325 mg dose), once daily and oral esomeprazole magnesium (40 mg, twice daily).
  acetylsalicylic acid: Given orally esomeprazole magnesium: Given orally placebo: Given orally
Period: Overall Study
Arm/Group | Arm I (Placebo, Esomeprazole Magnesium) | Arm II (Low-dose Aspirin, Placebo, Esomeprazole Magnesium) | Arm III (Higher-dose Aspirin, Palcebo, Esomeprazole Magnesium)
Started | 30 | 47 | 45
Completed | 29 | 42 | 43
Not Completed | 1 | 5 | 2
Not completed — Protocol Violation | 1 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Two patients from ARM II withdrew due to an inadequate number of biopsies and were not included in baseline measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Placebo, Esomeprazole Magnesium) | Arm II (Low-dose Aspirin, Placebo, Esomeprazole Magnesium) | Arm III (Higher-dose Aspirin, Palcebo, Esomeprazole Magnesium) | Total
Number analyzed (Participants) | 30 | 45 | 45 | 120
Age, Continuous [Median (Full Range); unit: years] | 61 [32 to 86] | 59 [34 to 81] | 59 [35 to 82] | 60 [32 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 7 | 19
  Male | 26 | 37 | 38 | 101
Region of Enrollment [Number; unit: participants]
  United States | 30 | 45 | 45 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Tissue Prostaglandin E2 (PGE2) Concentration as Determined From Barrett's Research Mucosal Biopsy Samples
Description: The mean tissue PGE2 is reported for each Arm.
Time Frame: Baseline to 30 days after completion of study treatment
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Arm I (Placebo, Esomeprazole Magnesium) | Arm II (Low-dose Aspirin, Placebo, Esomeprazole Magnesium) | Arm III (Higher-dose Aspirin, Palcebo, Esomeprazole Magnesium)
Number analyzed (Participants) | 29 | 42 | 43
pg/mL | -67.6 (229.68) [-745.2 to 454.7] | -123.9 (284) [-976.6 to 789] | -174.9 (263.62) [-1113.6 to 75.3]
Statistical Analysis 1: Comparison: Arm I (Placebo, Esomeprazole Magnesium) vs Arm II (Low-dose Aspirin, Placebo, Esomeprazole Magnesium); Test type: Superiority or Other; p = 0.0955, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (Placebo, Esomeprazole Magnesium) vs Arm III (Higher-dose Aspirin, Palcebo, Esomeprazole Magnesium); Test type: Superiority or Other; p = 0.0204, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Toxicity
Description: Toxicity is defined as adverse events that are classified as either possibly, probably, or definitely related to the interventional agent, graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. The number of patients reporting adverse events will be tabulated by grade.
Time Frame: Up to 30 days after completion of study treatment
Population: All 120 patients that took study medication were evaluable for this secondary endpoint.
Measure: Number; unit: participants
Arm/Group | Arm I (Placebo, Esomeprazole Magnesium) | Arm II (Low-dose Aspirin, Placebo, Esomeprazole Magnesium) | Arm III (Higher-dose Aspirin, Palcebo, Esomeprazole Magnesium)
Number analyzed (Participants) | 30 | 45 | 45
participants
  Grade 3 or Higher | 0 | 1 | 1
  Grade 4 or Higher | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (Placebo, Esomeprazole Magnesium) | Arm II (Low-dose Aspirin, Placebo, Esomeprazole Magnesium) | Arm III (Higher-dose Aspirin, Palcebo, Esomeprazole Magnesium)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/45 | 1/45
Other Adverse Events (participants affected / at risk) | 8/30 | 9/45 | 15/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Placebo, Esomeprazole Magnesium) (N=30) | Arm II (Low-dose Aspirin, Placebo, Esomeprazole Magnesium) (N=45) | Arm III (Higher-dose Aspirin, Palcebo, Esomeprazole Magnesium) (N=45)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Placebo, Esomeprazole Magnesium) (N=30) | Arm II (Low-dose Aspirin, Placebo, Esomeprazole Magnesium) (N=45) | Arm III (Higher-dose Aspirin, Palcebo, Esomeprazole Magnesium) (N=45)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (9)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (12) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (3) | 1 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (6) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less